CLINICAL TRIAL: NCT06487273
Title: Evaluation of the Impact of SIMEOX Airway Clearance Medical Device at Home, Combined With Remote Physiotherapy, on Quality of Life and Pulmonary Exacerbations in Patients With Non-cystic Fibrosis Bronchiectasis, Compared With Enhanced Standard of Care
Brief Title: Long-term Evaluation of the SIMEOX Device at Home in Non-cystic Fibrosis Bronchiectasis
Acronym: Home-BRAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Assist (Industry)
Collaborators: Icadom (Industry); Clinact (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A01095-40
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: Non-CF Bronchiectasis; Bronchial clearance

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, randomised according to modified Zelen method in two steps, controlled, multi-sites clinical investigation
  2 groups : comparison of SIMEOX + remote Physiotherapy + standard of care versus remote Physiotherapy + standard of care
Who Masked: Participant
Masking Description: modified Zelen method: participants in the control group will not be aware of another group using the SIMEOX -> only one group is blinded
  A blinded adjudication committee will review the outcome for one primary endpoint (exacerbations).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Remote Physiotherapy + standard of care
  Interventions: Other: Remote Physiotherapy
- SIMEOX (Experimental): SIMEOX device combined with Remote Physiotherapy + standard of care
  Interventions: Device: SIMEOX; Other: Remote Physiotherapy

INTERVENTIONS:
Device: SIMEOX — Use of the CE-marked SIMEOX medical device. No specific limitation of the number of use but recommendation to use it daily (and more if needed).
  Arms: SIMEOX
Other: Remote Physiotherapy — Remote Physiotherapy with physiotherapists, once a month for the first 3 months and once every 3 months after

SUMMARY:
Bronchiectasis is a chronic lung disease of multiple aetiologies characterised by permanent dilatation of the calibre of a territory of the bronchial tree with impaired mucociliary clearance. This alteration causes mucus retention, leading to infections and chronic bronchial inflammation. Respiratory physiotherapy is one of the cornerstones of the management of these patients, in particular to facilitate bronchial drainage. In patients with abundant bronchial secretions, it is recommended that bronchial drainage sessions be carried out on a daily or more frequent basis, which represents a very substantial burden in terms of care. In addition, access to respiratory physiotherapy is not always easy for patients due to geographical or time constraints or the availability of professionals. Moreover, few professionals are trained in this specific care for chronic lung diseases.

SIMEOX (Physio-Assist, France) is an innovative medical device (CE medical mark) for draining the bronchial tree. By means of a mouthpiece, this device generates a succession of very short intermittent negative air pressure pulses which disseminate a pneumatic vibratory signal in the patient's bronchial tree, modifying the rheological properties of the mucus, facilitating the mobilisation of secretions and assisting their transport towards the upper airways.

A recent pilot study demonstrated that the use of SIMEOX independently by the patient at home for 3 months, combined with remote Physiotherapy (1 session/2 weeks), provided a very satisfactory bronchial drainage solution for patients (satisfaction assessed at 9/10 by visual analogue scale), with an improvement in their quality of life and very good compliance with the device (median of 4.7 sessions/week).

This bronchial drainage strategy requires a long-term assessment.

Hypothesis: the use of SIMEOX independently by the patient at home could improve long-term quality of life and reduce the rate of pulmonary exacerbations in non-cystic fibrosis (non-CF) patients with bronchiectasis (bronchial dilatation) in comparison to Standard of Care (SoC).

DETAILED DESCRIPTION:
Two main objectives will be assessed simultaneously:

* To compare the effect of SIMEOX, combined with remote Physiotherapy, with enhanced SoC (SoC + Remote Physiotherapy), on the quality of life related to the respiratory problems of patients at mid term.
* To compare the effect of SIMEOX, combined with remote Physiotherapy with enhanced SoC (SoC + Remote Physiotherapy) on the rate of respiratory exacerbations at long term.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18 years
* Predominant diagnosis of Non CF bronchiectasis disease, excluding cystic fibrosis, confirmed by computed tomography (CT).
* Regular and chronic sputum production
* Clinically stable at inclusion

  * Defined by a delay of at least 4 weeks since the end of the last exacerbation according to the European consensus (Hill, European Respiratory Journal, 2017)
  * No change in disease-modifying treatment for 4 weeks.
* Having had at least two pulmonary exacerbations in the 12 months prior to inclusion and having required a change in specific treatment for these exacerbations.

Or Having had at least one pulmonary exacerbation in the 12 months prior to inclusion requiring hospitalisation.

* Considered by the investigator to be physically and psychologically able to use the device and carry out the procedures under study.
* Patient covered by a social security system, when applicable in the concerned country

Exclusion Criteria:

* Patients using one of the following motorised mechanical bronchial drainage devices at home at the time of inclusion:

  * SIMEOX,
  * an extra-thoracic high-frequency chest wall oscillation device (HFCWO) (The Vest,...)
  * intrapulmonary percussion ventilation (IPV)
* Patients who have been using a powered mechanical cough aid at home for less than a year at the time of inclusion:

  * a mechanical in-exsufflator (MI E) such as the Cough Assist
  * a pressure reducer such as the Alpha300
* Cystic fibrosis
* Predominant diagnosis of Chronic obstructive pulmonary disease (COPD) or asthma, traction bronchiectasis, bronchiectasis resulting from focal endobronchial lesion, sarcoidosis or active allergic bronchopulmonary aspergillosis.
* Active smoking
* Suspected (but undiagnosed) or unstabilised immune deficiency (at investigator's discretion)
* In the case of long-term immunosuppressive treatment, risk of discontinuation of this treatment during the study.
* Unstable cardiovascular pathologies (acute coronary syndrome, unstable angina pectoris, uncontrolled rhythm disorders, unstable heart failure)
* Haemodynamic instability
* Uncontrolled gastro-oesophageal reflux (persistence of symptoms despite treatment), at investigator's discretion.
* Acute pneumothorax or increased susceptibility to pneumothorax/pneumomediastinum
* Inability to cough vigorously and independently, at investigator's discretion
* Had a significant episode of haemoptysis in the 6 weeks prior to inclusion, at the discretion of the investigator
* Patient using an endotracheal tube, tracheostomy tube or daytime ventilation >16h with a mask
* Patients with neuromuscular disease and respiratory muscle weakness, at the discretion of the investigator
* Recent cardiothoracic surgery, including oesophageal surgery within 3 months of inclusion
* Severe acute lung injury or barotrauma within 3 months of inclusion
* Difficulty in evacuating secretions from the upper airways due to weakness of the respiratory muscles, or of the oropharyngeal or buccal musculature, at the discretion of the investigator
* Risk of airway aspiration, e.g. from tube feeding or recent meals, at investigator's discretion
* Inspiratory muscle weakness with inability to tolerate increased work of breathing, at investigator's discretion
* Severe restrictive disease (Forced Vital Capacity < 60% or Total Lung Capacity < 60% with complete plethysmography)
* Bullous emphysema
* Participation in other interventional clinical study in the month prior to inclusion or during the study period
* Patient unavailable or wishing to move to a region where the protocol is not present before the end of their participation
* Vulnerable people:

  * pregnant women (verified by a urine or blood human chorionic gonadotropin (HCG) test for all women wishing to participate in the protocol and of childbearing age, without contraception), breastfeeding mothers or women planning to become pregnant during the period of participation in the clinical investigation
  * a person deprived of liberty by judicial or administrative decision
  * a person subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life SGRQ at 6 months | Change from baseline at 6 months
  The change in the St George's Hospital Respiratory Questionnaire total quality of life score from baseline (inclusion) at 6 months of treatment, adjusted on the baseline score, with a comparison between the SIMEOX-treated group and the control group.
The annual rate of pulmonary exacerbations | Over the duration of the study (24 months in average)
  The annual rate of pulmonary exacerbations observed per patient per year compared between the SIMEOX-treated group and the control group over the duration of the study (24 months in average).

SECONDARY OUTCOMES:
Quality of life SGRQ at 12 months | Change from baseline at 12 months
  The change in total quality of life score measured by the St George's Respiratory Questionnaire from baseline at 12 months of treatment, adjusted for the baseline score, will be compared between the SIMEOX-treated group and the control group.
Quality of life SGRQ at 24 months | Change from baseline at 24 months
  The change in total quality of life score measured by the St George's Respiratory Questionnaire from baseline at 24 months of treatment, adjusted for the baseline score, will be compared between the SIMEOX-treated group and the control group.
3 domains of quality of life of the SGRQ at 6 months | Change from baseline at 6 months
  The change in scores of any of the 3 domains of quality of life of the St George's Respiratory Questionnaire from baseline at 6 months of treatment, adjusted for the score at inclusion, compared between the SIMEOX-treated group and the control group.
3 domains of quality of life of the SGRQ at 12 months | Change from baseline at 12 months
  The change in scores of any of the 3 domains of quality of life of the St George's Respiratory Questionnaire from baseline at 12 months of treatment, adjusted for the score at inclusion, compared between the SIMEOX-treated group and the control group.
3 domains of quality of life of the SGRQ at 24 months | Change from baseline at 24 months
  The change in scores of any of the 3 domains of quality of life of the St George's Respiratory Questionnaire from baseline at 24 months of treatment, adjusted for the score at inclusion, compared between the SIMEOX-treated group and the control group.
QoL-B questionnaire at 6 months | Change from baseline at 6 months
  The change in specific quality of life measured by the QoL-B questionnaire (8 domains) from baseline at 6 months of treatment, adjusted on the baseline score, compared between the SIMEOX-treated group and the control group
QoL-B questionnaire at 12 months | Change from baseline at 12 months
  The change in specific quality of life measured by the QoL-B questionnaire (8 domains) from baseline at 12 months of treatment, adjusted on the baseline score, compared between the SIMEOX-treated group and the control group
QoL-B questionnaire at 24 months | Change from baseline at 24 months
  The change in specific quality of life measured by the QoL-B questionnaire (8 domains) from baseline at 24 months of treatment, adjusted on the baseline score, compared between the SIMEOX-treated group and the control group
EQ5D-5L questionnaire at 6 months | Change from baseline at 6 months
  The change in global quality of life measured by the EuroQol 5 D descriptive system-5 Level questionnaire (EQ5D-5L) from baseline at 6 months of treatment, adjusted on the baseline score, compared between the SIMEOX-treated group and the control group.
EQ5D-5L questionnaire at 12 months | Change from baseline at 12 months
  The change in global quality of life measured by the EQ5D-5L questionnaire from baseline at 12 months of treatment, adjusted on the baseline score, compared between the SIMEOX-treated group and the control group.
EQ5D-5L questionnaire at 24 months | Change from baseline at 24 months
  The change in global quality of life measured by the EQ5D-5L questionnaire from baseline at 24 months of treatment, adjusted on the baseline score, compared between the SIMEOX-treated group and the control group.
CAAT questionnaire at 6 months | Change from baseline at 6 months
  The change in the perception of respiratory health measured by the Chronic Airways Assessment Test (CAAT) questionnaire from baseline at 6 months of treatment, adjusted on the baseline score, will be compared between the SIMEOX-treated group and the control group.
CAAT questionnaire at 12 months | Change from baseline at 12 months
  The change in the perception of respiratory health measured by the Chronic Airways Assessment Test (CAAT) questionnaire from baseline at 12 months of treatment, adjusted on the baseline score, will be compared between the SIMEOX-treated group and the control group.
CAAT questionnaire at 24 months | Change from baseline at 24 months
  The change in the perception of respiratory health measured by the Chronic Airways Assessment Test (CAAT) questionnaire from baseline at 24 months of treatment, adjusted on the baseline score, will be compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEV1 at 6 months | Change from inclusion at 6 months
  The change of the Forced expiratory volume in 1 second (FEV1) spirometry parameter of the respiratory function from inclusion at 6 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEV1 at 12 months | Change from inclusion at 12 months
  The change of the FEV1 spirometry parameter of the respiratory function from inclusion at 12 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEV1 at 24 months | Change from inclusion at 24 months
  The change of the FEV1 spirometry parameter of the respiratory function from inclusion at 24 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FVC at 6 months | Change from inclusion at 6 months
  The change of the Forced vital capacity (FVC) spirometry parameter of the respiratory function from inclusion at 6 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FVC at 12 months | Change from inclusion at 12 months
  The change of the FVC spirometry parameter of the respiratory function from inclusion at 12 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FVC at 24 months | Change from inclusion at 24 months
  The change of the FVC spirometry parameter of the respiratory function from inclusion at 24 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEV1/FVC at 6 months | Change from inclusion at 6 months
  The change of the FEV1/FVC spirometry parameter of the respiratory function from inclusion at 6 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEV1/FVC at 12 months | Change from inclusion at 12 months
  The change of the FEV1/FVC spirometry parameter of the respiratory function from inclusion at 12 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEV1/FVC at 24 months | Change from inclusion at 24 months
  The change of the FEV1/FVC spirometry parameter of the respiratory function from inclusion at 24 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEF 25-75% at 6 months | Change from inclusion at 6 months
  The change of the Forced mid-expiratory flow rate between 25% and 75% of the vital capacity (FEF 25-75%) spirometry parameter from inclusion at 6 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEF 25-75% at 12 months | Change from inclusion at 12 months
  The change of the FEF 25-75% spirometry parameter of the respiratory function from inclusion at 12 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
spirometry parameters : FEF 25-75% at 24 months | Change from inclusion at 24 months
  The change of the FEF 25-75% spirometry parameter of the respiratory function from inclusion at 24 months of treatment, adjusted on the baseline values, compared between the SIMEOX-treated group and the control group.
Time period before first exacerbation | Over the duration of the study (24 months in average)
  The time period, in days, between the date of randomisation and the start of the first respiratory exacerbation (as defined in the main co-criterion) compared between the SIMEOX-treated group and the control group
Rate of respiratory exacerbations with hospitalisation at 6 months | 6 months
  The rate of respiratory exacerbations (as defined in the main co-criterion) with hospitalisation observed per patient per year at 6 months of treatment, compared between the SIMEOX-treated group and the control group.
  Hospitalisations will be documented according to whether the patient is admitted in conventional care or intensive care/resuscitation.
Rate of respiratory exacerbations with hospitalisation at 12 months | 12 months
  The rate of respiratory exacerbations (as defined in the main co-criterion) with hospitalisation observed per patient per year at 12 months of treatment, compared between the SIMEOX-treated group and the control group.
  Hospitalisations will be documented according to whether the patient is admitted in conventional care or intensive care/resuscitation.
Rate of respiratory exacerbations with hospitalisation over the duration of the study | Over the duration of the study (24 months in average)
  The rate of respiratory exacerbations (as defined in the main co-criterion) with hospitalisation observed per patient per year over the duration of the study (24 months in average), compared between the SIMEOX-treated group and the control group.
  Hospitalisations will be documented according to whether the patient is admitted in conventional care or intensive care/resuscitation.
Rate of respiratory exacerbations without hospitalisation at 6 months | 6 months
  The rate of respiratory exacerbations (as defined in the main co-criterion) without hospitalisation observed per patient per year at 6 months of treatment, compared between the SIMEOX-treated group and the control group.
  Hospitalisations will be documented according to whether the patient is admitted in conventional care or intensive care/resuscitation.
Rate of respiratory exacerbations without hospitalisation at 12 months | 12 months
  The rate of respiratory exacerbations (as defined in the main co-criterion) without hospitalisation observed per patient per year at 12 months of treatment, compared between the SIMEOX-treated group and the control group.
  Hospitalisations will be documented according to whether the patient is admitted in conventional care or intensive care/resuscitation.
Rate of respiratory exacerbations without hospitalisation over the duration of the study | Over the duration of the study (24 months in average)
  The rate of respiratory exacerbations (as defined in the main co-criterion) without hospitalisation observed per patient per year over the duration of the study (24 months in average), compared between the SIMEOX-treated group and the control group.
  Hospitalisations will be documented according to whether the patient is admitted in conventional care or intensive care/resuscitation.
Proportion of patients with 2 or more exacerbations at 6 months | 6 months
  The proportion of patients with 2 or more exacerbations observed at 6 months of treatment will be compared between the SIMEOX-treated group and the control group.
Proportion of patients with 2 or more exacerbations at 12 months | 12 months
  The proportion of patients with 2 or more exacerbations observed at 12 months of treatment will be compared between the SIMEOX-treated group and the control group.
Proportion of patients with 2 or more exacerbations over the duration of the study | Over the duration of the study (24 months in average)
  The proportion of patients with 2 or more exacerbations observed over the duration of the study will be compared between the SIMEOX-treated group and the control group.
Proportion of patients with at least one hospitalisation for exacerbations at 6 months | 6 months
  The proportion of patients with at least one hospitalisation for exacerbations observed at 6 months of treatment will be compared between the SIMEOX-treated group and the control group.
Proportion of patients with at least one hospitalisation for exacerbations at 12 months | 12 months
  The proportion of patients with at least one hospitalisation for exacerbations observed at 12 months of treatment will be compared between the SIMEOX-treated group and the control group.
Proportion of patients with at least one hospitalisation for exacerbations over the duration of the study | Over the duration of the study (24 months in average)
  The proportion of patients with at least one hospitalisation for exacerbations observed over the duration of the study will be compared between the SIMEOX-treated group and the control group.
Duration of hospitalisation for exacerbations at 6 months | 6 months
  The duration of hospitalisation for exacerbations observed at 6 months of treatment will be compared between the SIMEOX-treated group and the control group.
Duration of hospitalisation for exacerbations at 12 months | 12 months
  The duration of hospitalisation for exacerbations observed at 12 months of treatment will be compared between the SIMEOX-treated group and the control group.
Duration of hospitalisation for exacerbations over the duration of the study | Over the duration of the study (24 months in average)
  The duration of hospitalisation for exacerbations observed over the duration of the study will be compared between the SIMEOX-treated group and the control group.
The percentage of responder / non-responder patients at 12 months | 12 months
  The percentage of responder / non-responder patients from inclusion at 12 months of treatment will be assessed by:
  * a change in St George's Hospital Respiratory Questionnaire (SGRQ) total quality of life score greater than minimal clinically important difference (MCID) (> or equal to 4 points),
  and/or
  * the absence of pulmonary exacerbation during this period.
  Patients belonging to the other categories (SGRQ variation < 4 and presence of one or more pulmonary exacerbations) will be classified as non-responders at 12 months of treatment.
The percentage of responder / non-responder patients at 24 months | 24 months
  The percentage of responder / non-responder patients patients from inclusion at 24 months of treatment, will be assessed by:
  * a change in St George's Hospital Respiratory Questionnaire (SGRQ) total quality of life score greater than MCID (> or equal to 4 points),
  and/or
  * the absence of pulmonary exacerbation during this period.
  Patients belonging to the other categories (SGRQ variation < 4 and presence of one or more pulmonary exacerbations) will be classified as non-responders at 24 months of treatment.
Average number of sessions | Over the duration of the study (24 months in average)
  Changes in adherence to the SIMEOX device will be described by the average number of sessions performed by the patient over the entire follow-up period and for each month/quarter of participation
Proportion of compliant patients | Over the duration of the study (24 months in average)
  The proportion of compliant patients will be evaluated by the percentage of patients having performed 3 sessions or more per week over the entire follow-up period and for each quarter (SIMEOX group only).
Number of adverse events | Over the duration of the study (24 months in average)
  Safety of use will be assessed by the number of adverse events related to the procedure for using the medical device or to the medical device itself over the course of the study (24 months in average). These will be counted and qualified as serious or non-serious.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Leroy, MD, Principal Investigator — CHU NICE
Locations (43):
- France (41):
  - CH Abbeville, Abbeville
  - CH Aix en Provence, Aix-en-Provence
  - CH Albi, Albi
  - Clinique Victor Pauchet, Amiens
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CH Annecy, Annecy
  - Clinique Aressy, Aressy
  - CHRU Brest, Brest
  - CH Cotentin, Cherbourg
  - CH Compiègne-Noyon, Compiègne
  - CH Alpes-Léman, Contamine-sur-Arve
  - CHI Créteil, Créteil
  - CFR Dieulefit, Dieulefit
  - CHU Grenoble-Alpes, Grenoble
  - HCL - centre de Hyères, Hyères
  - Groupe Hospitalier La Rochelle - Ré-Aunis, La Rochelle
  - Hôpital Bicêtre (AP-HP), Le Kremlin-Bicêtre
  - CH Le Puy-en-Velay, Le Puy-en-Velay
  - CH Libourne, Libourne
  - CHU Limoges, Limoges
  - HCL- Hôpital Croix-Rousse, Lyon
  - Hôpital Européen de Marseille, Marseille
  - Groupe Hospitalier du Havre, Montivilliers
  - Montpellier Hospital Center, Montpellier
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - Hôpital Cochin (AP-HP), Paris
  - CH Pau, Pau
  - CH Perpignan, Perpignan
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - Fondation Ildys, Roscoff
  - CHU Rouen, Rouen
  - CH St Quentin, Saint-Quentin
  - Hôpital Foch, Suresnes
  - CH Tarbes Lourdes, Tarbes
  - CHU Toulouse, Toulouse
  - CH Troyes, Troyes
  - CH Bretagne Atlantique, Vannes
- Reunion (2):
  - CHU La Réunion Félix Guyon, Saint-Denis
  - CHU La Réunion Sud, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamidfar R, Murris-Espin M, Mahot M, Abouly R, Gauchez H, Jacques S, Joffray E, Arnol N, Morin L, Leroy S, Borel JC. Feasibility of home initiation of an airway clearance device (SIMEOX) by telecare in people with non-cystic fibrosis bronchiectasis: a pilot study. BMJ Open Respir Res. 2023 Jul;10(1):e001722. doi: 10.1136/bmjresp-2023-001722. PMID 37524523